CLINICAL TRIAL: NCT05471011
Title: Multi-Dimensional Outcome Prediction Algorithm for Hospitalized COVID-19 Patients
Brief Title: COVID-19 Outcome Prediction Algorithm
Acronym: COPA
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Olive View-UCLA Education & Research Institute (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Atlanta VA Medical Center (U.S. Federal Agency); Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mario C. Deng, Professor of Medicine, University of California, Los Angeles
Other Study IDs: 1R01AI159946-01A1 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Post Acute Sequelae of COVID-19; Long COVID; Organ Dysfunction Syndrome, Multiple; Frailty Syndrome
Keywords: outcome prediction; systems biology; multiomics; algorithm; veterans; high-risk populations
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Multiple Organ Failure; Frailty | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- civilian
  Interventions: Other: Blood and nasal swab sampling
- Veteran
  Interventions: Other: Blood and nasal swab sampling

INTERVENTIONS:
Other: Blood and nasal swab sampling — Blood and nasal swab sampling

SUMMARY:
Severe acute respiratory syndrome coronavirus 2-mediated coronavirus disease (COVID-19) is an evolutionarily unprecedented natural experiment that causes major changes to the host immune system. We propose to develop a test that accurately predicts short- and long-term (within one-year) outcomes in hospitalized COVID-19 patients broadly reflecting US demographics who are at increased risk of adverse outcomes from COVID-19 using both clinical and molecular data. We will enroll patients from a hospitalized civilian population in one of the country's largest metropolitan areas and a representative National Veteran's population.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-mediated coronavirus disease (COVID-19) is an evolutionarily unprecedented natural experiment that causes major changes to the host immune system. Several high risk COVID-19 populations have been identified. Older adults, males, persons of color, and those with certain underlying health conditions (e.g., diabetes mellitus, obesity, etc.) are at higher risk for severe disease from COVID-19. While it is too soon to fully understand the impact of COVID-19 on overall health and well-being, there are already several reports of significant sequelae, which appear to correlate with disease severity. There is a clear and urgent need to develop prediction tests for adverse short- and long-term outcomes, especially for high-risk COVID-19 populations. We hypothesize that complementary multi-dimensional information gathered near the time of symptom onset can be used to predict new onset or worsening frailty, organ dysfunction and death within one year after COVID-19 onset. A single parameter provides limited information and is incapable of adequately characterizing the complex biological responses in symptomatic COVID-19 to predict outcome. Since they were designed for other illnesses, it is unlikely that existing clinical tools, such as respiratory, cardiovascular, and other organ function assessment scores, will precisely assess the long-term prognosis of this novel disease. Our extensive experience in biomarker development suggests that integrating molecular and clinical data increases prediction accuracy of long-term outcomes. We have chosen to test our hypothesis in a population reflecting US-demographics that is at increased risk of adverse outcomes from COVID-19. We will enroll patients, broadly reflecting US demographics, from a hospitalized civilian population in one of the country's largest metropolitan areas and a representative National Veteran's population. We anticipate that a prediction test that performs well in this hospitalized patient group will: help guide triaging and treatment decisions and, therefore, reduce morbidity and mortality rates, enhance patient quality of life, and improve healthcare cost-effectiveness. More accurate prognostic information will also assist clinicians in framing goals of care discussions in situations of likely futility and assist patients and families in this decision-making process. Finally, it will provide a logical means for allocating resources in short supply, such as ventilators or therapeutics with limited availability.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic COVID-19 infection with hospital admission
* Age 18 and above
* Informed consent

Exclusion Criteria:

* Absence of symptomatic COVID-19 infection with hospital admission
* Age 17 or below
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic COVID-19 infected civilians and symptomatic COVID-19 infected veterans
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
New onset or worsening frailty, single organ dysfunction, multi-organ dysfunction, and death within one year | From hospital admission to one year
  The primary outcome clinical composite endpoints that include new onset or worsening frailty, single organ dysfunction, multi organ dysfunction, and death within one year will include a follow-up period of time of at least 52 weeks after initial enrollment encounter. The assessment of time to event (outcome events will include various frailty measurement tools including short physical performance battery, laboratory test-based organ function assessment measures, and survival status as per publicly-accessible databases) will consist of calculating the time difference between first outcome event and baseline encounter date.

SECONDARY OUTCOMES:
New onset or worsening frailty, single organ dysfunction, multi-organ dysfunction, and death at time of discharge | From hospital admission to time of discharge
  The secondary outcome clinical composite endpoints that include new onset or worsening frailty, single organ dysfunction, multi organ dysfunction, and death within the time from initial encounter to the time of discharge will include a follow-up period consisting of the time from initial enrollment encounter to the time of discharge. The assessment of time to event (outcome events will include various frailty measurement tools including short physical performance battery, laboratory test-based organ function assessment measures, and survival status as per publicly-accessible databases) will consist of calculating the time difference between first outcome event and baseline encounter date.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Olive View-UCLA Education & Research Institute, Sylmar, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Atlanta VA Medical Center, Decatur, Georgia
  - Bronx VA Medical Center, The Bronx, New York
  - Michael E. DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
After our data is cleaned, quality checked, and analyzed, we will make the data available to the general research community. Data collected in this proposal will be submitted to the appropriate public databases (e.g. Gene Expression Omnibus), along with complete documentation to enable efficient use of the data by the general research community. Cumulative datasets will be submitted on a regular basis in a timely manner. All data made available for public use will be de-identified data, i.e., stripped of private, protected health information that could be used to deduce the identity of individual subjects, in compliance with the HIPPA Privacy Rule. The study will be registered in the database of Genotypes and Phenotypes and the following data and information will be shared through the Sequence Read Archive and Gene Expression Omnibus.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available following the completion of the study and will be available indefinitely.
Access Criteria: COPA Study website to be determined

REFERENCES:
- [Background] Deng MC. Multi-dimensional COVID-19 short- and long-term outcome prediction algorithm. Expert Rev Precis Med Drug Dev. 2020;5(4):239-242. doi: 10.1080/23808993.2020.1785286. Epub 2020 Jun 24. No abstract available. PMID 33283045

DOCUMENTS (1):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT05471011/Prot_000.pdf